CLINICAL TRIAL: NCT06899789
Title: Long-term Follow-up of Checkpoint Inhibitors-induced Ileo-colitis
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Marco Vincenzo Lenti, Prof, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: ICIC-ECCO
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-02

CONDITIONS: Immune Checkpoint Inhibitors-induced Colitis; Advanced Melanoma Skin Cancer, Non-small Cell Lung Carcinoma, Kidney Adenocarcinoma; Ileo-colitis; Immune Mediated-colitis
Keywords: Immune checkpoint inhibitors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Newly diagnosed of CIC patients, with a proven endoscopic and histological diagnosis: The study will include all patients developing colitis (diagnosed with endoscopy and/or histological examination) after at least one administration of a checkpoint inhibitor therapy for advanced cancer. Patients with a previous diagnosis of IBD (before cancer onset or before immunotherapy beginning) will be excluded, as well as patients with a previous diagnosis of other forms of colitis (other than IBD).

SUMMARY:
This is a multicentric, observational study, including all European centres willing to take part. The multicentre nature is necessary for enhancing the generalisability of our results, and due to the rarity of this condition. The study is observational including both retrospective and newly diagnosed cases of CIC with an endoscopically/histologically-proven diagnosis. Detailed characteristics will be collected, with the aim of classifying the disorders from a clinical, endoscopic, and pathological point of view. Age, sex, localisation, and histology of tumour, stage of tumour, oncological response to immune checkpoint inhibitors-induced colitis, colonoscopy, histology, inflammatory parameters, and clinical manifestations will be assessed for each patient, as well as therapy and outcome.

The study will consist of 2 part: the first one will be retrospective, while the second one will be prospective al will include all incident patients diagnosed with CIC during the enrolment period.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* patients able to provide informed consent or who have already given leave of use of their data for research in the retrospective part; waiving of the informed consent may be applied if national regulations allow to do so;
* patients who have undergone at least one cycle of immune checkpoint inhibitors before the onset of intestinal symptoms;
* patients with at least one colonoscopy showing macroscopical and/or histological colitis after commencement of immune checkpoint inhibitors therapy; for retrospective patients only, a follow-up of at least 12 months, unless death occurred before.

Exclusion Criteria:

* Evidence of colitis/inflammatory bowel disease prior to checkpoint inhibitors administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a histologically proven CIC or enterocolitis. Any cancer patient who is started on any available immune check-point inhibitor and developing CIC/enterocolitis will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the rate of clinical remission defined as symptoms CTCAE grade 1 or less within 12 months after CIC diagnosis (at the last evaluation available when death occurs or at one year from diagnosis). | After baseline evaluation at the time of immune CIC diagnosis and four other evaluations after 3, 6, 9, and 12 months or until death if death occurred in the first 12 months.
  The rate of remission at 12 months will be estimated together with its 95% exact binomial 95% CI. The association of a series of predefined non-collinear baseline covariates and remission will be assessed using multivariable logistic regression. Huber-White robust standard errors will be computed to account for intra-centre correlation of measures. In case of death prior to the 12-month assessment, the last available measure will be used. A sensitivity analysis of the primary endpoint may be performed using multiple imputation of the primary endpoint for those patients who do not reach the 12 months assessment due to death or loss to follow-up. The following covariates will be considered: mild colitis vs those who need immunosuppressants, age >70 years, female sex, BMI>25, number of comorbidities, type of cancer (localisation, histology, and stage), type of ICI. A sensitivity analysis of the primary endpoint will be performed as described above with death considered as a failure.

CONTACTS AND LOCATIONS:
Locations (1):
- SC Medicina Generale 1, Fondazione IRCCS Policlinico san Matteo, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No